CLINICAL TRIAL: NCT03385473
Title: Individualized Antiretroviral Therapy: Impact of Pharmacogenetic and Therapeutic Drug Monitoring in the Safety and Efficacy of First Line Antiretroviral Therapy in Patients With HIV Infection
Brief Title: Individualized Antiretroviral Therapy
Acronym: IAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Waldo Horacio Belloso, MD, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1901
Record Dates: First submitted 2017-11-15; First posted 2017-12-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2020-07

CONDITIONS: Pharmacogenetics; HIV; Drug Monitoring
MeSH Terms: interventions — Drug Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacological Adequation (PA) (Active Comparator): Pharmacological adequation based on the Pharmacogenomic Index and therapeutic drug monitoring results.
  Interventions: Genetic: Pharmacogenomic index; Diagnostic Test: Therapeutic drug monitoring
- Standard of Care (SOC) (No Intervention): Without pharmacological adequation

INTERVENTIONS:
Genetic: Pharmacogenomic index — All patients will have a blood sample drawn at randomization visits for PG analysis. For patients in the PA arm, the sample will be processed immediately to obtain the PG results and the subsequent index within 10 days. As soon as the results are available, the project team will contact the attending physician to propose the dosing adequation according to the pharmacogenomic index. PG analysis will be performed once for each patient.
  Other Names: Diagnostic test
  Arms: Pharmacological Adequation (PA)
Diagnostic Test: Therapeutic drug monitoring — The patients included in the Pharmacological Adequation arm will have a TDM according to this schedule: day +14 (±3), +28 (±3), and +168 (±3). If there is an abnormal value (out of the therapeutic range), we will proceed to adjust the prescription.
  Other Names: TDM
  Arms: Pharmacological Adequation (PA)

SUMMARY:
The efficacy and safety of antiretroviral therapy and the damage caused by chronic inflammation in the presence of the virus has recently lead to the consideration of initiating antiretroviral therapy earlier than what is required to prevent opportunistic diseases.

Although there may be subtle differences, all recommended antiretroviral combinations for first-line therapy are considered equally effective. Nevertheless, treatment success requires high levels of adherence, which is linked to tolerability and the minimization of adverse effects.

The genes coding the enzymes that are involved in the antiretroviral clearance pathways and the transmembrane transport of drugs are known. These genetic variations can determine the interindividual variations in plasma concentration with the same doses. Both pharmacogenomics (PG) and therapeutic drug monitoring (TDM) may contribute to the individualization of therapy in different chronic conditions through dosing optimization and are associated with a lower risk of concentration-dependent toxicity and potentially greater efficacy. The use of these strategies in the context of antiretroviral therapy is in early stage of development.

Following, our main hypothesis is that PG + TDM dose adjustment of efavirenz or atazanavir in the initial antiretroviral treatment of naive patients with HIV infection is non-inferior in terms of efficacy, has improved safety, and shows a better cost/effectiveness profile than the standard approach with non adjusted doses.

To evaluate our hypothesis we developed this multicenter randomized clinical trial, where patients from 4 clinical sites in Buenos Aires will be included in the protocol and randomized to standard of care (SOC) or pharmacological adaptation (PA) -PA: PG + TDM. For the pharmacogenomics determination, we developed a multiplex approach including main polymorphisms of CYP2B6, CYP2A6, CYP3A4 y ABCB1 for efavirenz; and UGT1A1, ABCB1 and CYP3A4 for atazanavir. Drug plasma levels will be analyzed with ultra-performance liquid chromatography (UPLC).

The main outcomes are to establish the usefulness of PG and TDM in determining the efficacy, safety and cost/effectiveness of a first-line antiretroviral therapy containing either efavirenz or atazanavir in patients with HIV infection who have not received prior antiretroviral therapy.

DETAILED DESCRIPTION:
I) General Objectives To establish the overall impact of pharmacogenomic (PG) analysis and therapeutic drug monitoring (TDM) for the selection of the proper dose of efavirenz or atazanavir in patients with an HIV infection who have not received prior antiretroviral treatment.

II) Specific objectives and working hypothesis Establish the usefulness of PG and TDM in determining the efficacy, safety and cost/effectiveness of a first-line antiretroviral therapy containing either efavirenz or atazanavir in patients with HIV infection who have not received prior antiretroviral therapy.

II b. Working Hypothesis Pharmacogenomic analysis and therapeutic drug monitoring dose adjustment of efavirenz or atazanavir in the initial antiretroviral treatment of naive patients with HIV infection is non-inferior in terms of efficacy, has improved safety, and shows a better cost/effectiveness profile than the standard approach without dose adjustment.

III) Background III a. Introduction Combination antiretroviral therapy has modified the natural history of HIV infection in an unprecedented manner in medical history.

Today, the life expectancy of people with a chronic retroviral infection and access to treatment resembles that of the general population. The efficacy and safety of antiretroviral therapy and the damage caused by chronic inflammation in the presence of the virus has recently lead to the consideration of initiating antiretroviral therapy earlier.

Although there may be subtle differences in the effectiveness and speed of viral load reduction among the currently available drugs, all recommended antiretroviral combinations for first-line therapy are considered equally effective. Nevertheless, antiretroviral treatments present difficulties. Beyond the cost, which is covered by national health programs in most countries that provide medications, treatment success requires high levels of adherence, which is linked to tolerability and the minimization of adverse effects.

Selecting an adequate drug should not only be restricted to the selection of the components of the therapy, but it should also include the dosing and administration recommendations for each drug, aspects that are currently managed in a standard and uniform way that does not account for the particular characteristics of each patient.

Appearing in therapeutics to combat a pandemic, most antiretroviral drugs have been commercialized with the minimum information required to prove the efficacy and safety of the drugs. Following, much information is still being gathered in the post-marketing stage. In addition, the original developmental studies toward the approval of atazanavir were performed without ritonavir boosting in naive patients with HIV infection.

The metabolic pathways that participate in antiretroviral clearance are well defined, and the variations in the genes coding the enzymes that are involved in these pathways and the trans-membrane transport of drugs are known. Even considering these variations, a clear dose-response relationship defining reference therapeutic ranges has been established for many of these drugs.

Both pharmacogenomic and therapeutic drug monitoring may contribute to the individualization of therapy in different chronic conditions through dosing optimization and are associated with a lower risk of concentration-dependent toxicity and potentially greater efficacy.

III b. Applicability In most Latin American countries, approximately two-thirds of the first-line antiretroviral combinations include two nucleos(t)ides reverse transcriptase inhibitors and a non-nucleoside reverse transcriptase inhibitor, primarily efavirenz.

The other patients are treated with a protease inhibitor-based regimen that primarily includes atazanavir or lopinavir boosted with ritonavir.

The efficacy of antiretroviral treatments is high, and the therapeutic objective is to achieve an undetectable viral load in all patients. However, unpredictable circumstances related to tolerability and safety could lead to the modification or interruption of a significant proportion of initial antiretroviral combinations (between 20% and up to 45%).

Guidance based upon PG and TDM may aid in identifying patients with a higher risk of intolerance or toxicity and allow both initial dosing and subsequent posology adjustments to successfully maintain the utility of the drugs and minimize undesired effects.

III c. Genetic polymorphisms PG is the study of genetic variations related to individual drug responses. The variability in the expression of transporters, metabolizing enzymes and receptors is multifactorial but depends primarily on genetic factors.

There are different genetic variants among these hereditary factors, which may involve extensive portions of the cellular DNA. However the most frequent variations are single nucleotide polymorphisms (SNPs).

Genes that encode transporters, metabolizing enzymes or drug receptors may show different allelic variants that could impact the expression of the corresponding protein products.The study of these polymorphisms might predict the behavior of a specific pharmacologic process, and polymorphisms could be used to characterize patients. For example, patients could be characterized as slow or ultra-rapid metabolizers with respect to biotransformation enzymes. Modifying the dose or the dosing interval to obtain a desirable plasma concentration range of a drug is the major goal of an individualized prescription model.

For the vast majority of drugs, genotypic analysis of one metabolizing enzyme is not sufficient to characterize the complete genetic variability of a patient.In the near future, studies of potential polymorphisms in the genes of transporters and receptors will provide a better understanding of the pharmacogenomic impact of drug selection in a targeted therapeutic model. For most therapeutic areas in the meantime, current knowledge allows for a pharmacogenomic approach focused on the avoiding toxicity of drugs.

IV) Hypothesis and general methodology IV a. Introduction Currently available first-line antiretroviral treatment is usually administered in fixed doses without considering the pharmacokinetic particularities of different adult patients. The possibility of a useful tool that may help in the identification of these individual characteristics may allow a dosing adequation that is beneficial from both the safety and the economic perspectives.

In this sense, a combination of PG and TDM may allow a safe reduction in the efavirenz dose or the administration of atazanavir without booster in selected patients.

There are a number of publications regarding the potentially safe dose reduction of efavirenz and the use of atazanavir without ritonavir boosting in some patients both in case series and in multi-center cohorts, providing additional support for a prospective clinical trial.

IV b. Variables and tests As primary components of first-line antiretroviral combinations, therapeutic individualization will be focused on efavirenz and atazanavir. This decision is based upon two aspects: efavirenz and atazanavir constitute the most frequently used drugs in conjunction with nucleoside analogs, and in cohort studies, these drugs have been most clearly identified to be compromised by discontinuations resulting from genetic-related toxicities.

PG for Efavirenz: Polymorphisms of CYP2B6 (rs3745274), CYP2A6 (rs28399433/rs8192726), CYP3A4, (rs4646437), CYP3A4*1B and ABCB1 (rs1045642). For atazanavir: Polymorphisms of UGT1A1 (rs8175347), ABCB1 (rs10456542),polymorphisms of the steroid and xenobiotic receptor NR1 2 (rs2472677) TDM for Efavirenz (EFV) and Atazanavir (ATV): UPLC with diode arrangement and mass/mass detection.

V) Research Design and Methods A randomized prospective clinical study will be performed to evaluate the field utility of the therapeutic adjustment based on PG and TDM.

The objective population will be naive HIV-positive patients in whom starting antiretroviral treatment is warranted according to the attending physician's criteria and current antiretroviral treatment local guidelines, and efavirenz or atazanavir will be included in the therapeutic combination.

Candidates from five centers in Argentina will be invited to participate in this study through an informed consent process, after which patients will be randomized into one of the following arms:

* Standard of Care (SOC): without pharmacological adequation
* With Pharmacological Adequation (PA):based on the PG Index and TDM results Randomization will be performed using a random number sequence with restricted access with each new patient incorporation, fulfilling both components of the randomization process (random assignment and allocation concealment)

Follow up:

Patients included in the study will initiate their antiretroviral combination scheme within 2 weeks of enrollment.

All patients will have a blood sample drawn at randomization visits for PG analysis. For all patients included in the PA arm, the sample will be processed immediately, with the objective of obtaining the PG results and the subsequent index within 10 days. As soon as the results are available, one member of the project team will contact the attending physician to propose the corresponding dosing adjustment, which should be documented in the patient´s chart. PG analysis will be performed once for each patient.

The samples obtained from the patients in the SOC group will be stored after DNA extraction.

A viral genotyping test before treatment initiation will be performed at the discretion of the physician.

The patients included in the PA arm will have a TDM according to this schedule: day +14 (±3), +28 (±3), and +168 (±3). If there is an abnormal value (out of the therapeutic range), we will proceed to adjust the prescription according to the following recommendations:

Table 2. Drug dose adjustment according to the TDM results Antiretroviral drug Result Change in prescription Efavirenz: If above therapeutic range, reduce dose to 200 mg/d Efavirenz: If below therapeutic range, increase dose to 800 mg mg/d or change prescription to another drug Atazanavir: If above therapeutic range stop ritonavir or consider changing drug prescription Atazanavir: If below therapeutic range add ritonavir or consider changing drug prescription After the modification in dosing, a new TDM determination will be performed within a week.

All enrolled patients will be followed for one year. The efficacy/safety analysis of the interventions will be performed after 48 weeks.

After the initial visit and the initiation of antiretroviral treatment, patients will have 3 visits within one year. During each visit, we will perform a physical exam and a medical interview focusing on adverse events and the quality of life using a questionnaire.

Quality of life will be assessed using a validated questionnaire, FAHI (Functional Assessment of Human Immunodeficiency Virus Infection).

-Follow up schedule (both arms) Patient follow-up will be performed in accord with the standard of care for these patients with HIV viral load and CD4+ lymphocyte determinations every 4 months (±1 month). Because the results of the HIV viral load determination are part of the efficacy outcome of the study, the extraction/processing fee will be fully covered by the protocol, similar to the management of the TDM and PG determinations.

Medications Provided that the beginning of treatment and the selection of the therapeutic plan are chosen by the patient's physician and because the aim of the study is to evaluate the therapeutic plan, these drugs will be provided by the usual free-of-charge local delivery system. This project will not incur any additional costs, and is expected to provide economic savings to the health system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diagnosis of chronic HIV infection confirmed by Western blot and / or HIV viral load
* Patients in whom (according to the judgment of the treating physician) antiretroviral therapy should be initiated and this treatment will be a regimen based on Efavirenz or Atazanavir.
* Availability of a baseline genotyping test confirming the absence of primary resistance for the selected drugs.
* Signature of the informed Consent Form

Exclusion Criteria:

* Patients who remain untreated or those treated with a regimen that does not include efavirenz or atazanavir
* Lack of understanding of the study characteristics or rejection to have samples taken for the pharmacological studies.
* Patients who are not expected to continue their follow-up at the research center for at least one year
* Patients with coinfections or comorbidities that prevent a dose adjustment of efavirenz or atazanavir based on pharmacological parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementation of a multicenter study to analyze pharmacological adequation and therapeutic drug monitoring of efavirenz or atazanavir in the initial antiretroviral treatment of naive patients with HIV infection | 48 Weeks
  Number of days between obtention of study samples and availability of test results (turnaround time)

SECONDARY OUTCOMES:
Frequency of adverse events | 48 Weeks
  Pharmacological Adequation arm of efavirenz or atazanavir in the initial antiretroviral treatment of naive patients with HIV infection will show reduced frequency of adverse events when compared with the Standard Prescription arm.
Efficacy of antiretroviral treatment | 48 weeks
  Pharmacological Adequation arm of efavirenz or atazanavir performs equally to the standard of care arm. Viral load at 48 weeks aimed to be non inferior between arms, analyzed through FDA-recommended Snapshot approach.
Cost/effectiveness compared in both arms | 48 Weeks
  Pharmacological Adequation arm of efavirenz or atazanavir in the initial antiretroviral treatment of naive patients with HIV infection shows a better cost/effectiveness profile than the standard of care approach. (Direct Cost analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Waldo H Belloso, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires - Infectious Diseases Section, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided